CLINICAL TRIAL: NCT04801017
Title: A Double Blind, Randomized, Placebo Controlled, Multi Center Study of OT-101 in Hospitalized COVID-19 Subjects
Brief Title: A Study to Evaluate the Safety and Efficacy of OT-101+Artemisinin in Hospitalized COVID-19 Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oncotelic Inc. (Industry)
Responsible Party: Sponsor
Organization: Mateon Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C002 2020 01
Record Dates: First submitted 2021-03-01; First posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Trabedersen; artemisinin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OT-101 + Artemisinin + Standard of Care (Experimental): OT-101 - Days 1 to 7: 140 mg/m2 daily intravenous (i.v.) infusion for 7 continuous days.
  Artemisinin: Days 1 to 5: 500 mg per day for 5 days by oral
  Interventions: Drug: OT-101; Drug: Artemisinin
- Placebo + Artemisinin + Standard of Care (Placebo Comparator): Artemisinin: Days 1 to 5: 500 mg per day for 5 days by oral
  Interventions: Drug: Artemisinin; Drug: Placebo

INTERVENTIONS:
Drug: OT-101 — TGF β2 specific synthetic 18 mer phosphorothioate antisense oligodeoxynucleotide
  Other Names: Trabedersen
  Arms: OT-101 + Artemisinin + Standard of Care
Drug: Artemisinin — Herbal Supplement/ Purified extract from Artemisia
  Other Names: ArtiVeda
Drug: Placebo — 0.9% sodium chloride injection
  Other Names: Normal saline
  Arms: Placebo + Artemisinin + Standard of Care

SUMMARY:
Primary Objective is to evaluate the safety and efficacy of OT-101+Artemisinin when used in combination with standard of care (SoC) in hospitalized COVID 19 subjects versus SoC+ Artemisinin+Placebo.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled study to evaluate the efficacy, safety and tolerability of OT-101+Artemisinin when used in combination with SoC in hospitalized subjects with severe COVID 19. Written informed consent must be obtained from all subjects or their legally authorized representative (LAR) during screening (up to Day 3 prior to dosing) and prior to study related procedures being performed. Following completion of all screening assessments and meeting of eligibility criteria, subjects will be enrolled and randomized on Day 1 to either receive OT-101+Artemisinin or placebo+Artemisinin in a 2:1 ratio for 7 days in combination with SoC therapy per local SoC policies, followed to Day 28.

Subjects: includes subjects with severe COVID 19 (WHO COVID 19 Clinical Improvement Ordinal Scale 5 - non-invasive ventilation or high flow oxygen, or 6 - intubation and mechanical ventilation) at screening.

Subjects will undergo assessment during hospitalization or could discontinue their treatment with OT 101 or placebo during the 7 day infusion period or any time later during the study. All subjects will be closely monitored for adverse events (AEs) from signing the informed consent form (ICF) for at least 21 days after the final dose of study treatment (until Day 28). Standard of care treatment may continue as clinically indicated (after the 7 day dosing completion) as per local institutional guidelines. If subjects are discharged after Day 7 (after completing dosing), post discharge assessments can be done either at home (home health visit) or at the site. For subjects who are discharged before Day 28 or who withdraw from the study early will have follow up phone calls or will be followed up at site or a home visit to collect safety data until End of Study on Day 28. On days of laboratory assessments, discharged subjects may have a home visit.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized adult male or non-pregnant, non-lactating female subjects (between 18 and 80 years), with SARS-CoV-2 (previously known as 2019-nCoV) infection that is documented by authorized diagnostic PCR test. A rapid PCR test could also be used. Confirmation that subject has COVID-19 within the last 2 weeks prior to randomization.
2. Meeting WHO COVID 19 Clinical Improvement Ordinal Scale Criteria 5 (non-invasive mechanical ventilation or high-flow oxygen) or Criteria 6 (intubation and mechanical ventilation).
3. O2 sat <= 93%
4. Male subjects and female subjects of childbearing potential must agree to use protocol specified methods of contraception.
5. Female subjects of childbearing potential and women of non childbearing potential (defined as at least 2 years postmenopausal or permanently sterilized women [bilateral tubal ligation, bilateral ovariectomy, or hysterectomy]) must have a negative serum pregnancy test at screening or pretreatment on Day 1.
6. The subject or a LAR has provided written informed consent.
7. The subject or the LAR is aware of the investigational nature of this study and willing to comply with protocol treatments, and other evaluations listed in the ICF.

Exclusion Criteria:

1. Participation in any other clinical trial of an experimental treatment for COVID-19 or participation in another interventional clinical trial, including an expanded access trial.
2. Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS CoV 2 infection <24 hours prior to study drug dosing except for remdesivir.
3. Uncontrolled hypertension (systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), unstable angina, congestive heart failure of any New York Respiratory Association classification, serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia), or history of myocardial infarction within 12 months of enrollment.
4. Hypotension requiring vasoactive peptides, such as dopamine, norepinephrine, epinephrine, or dobutamine.
5. Renal function impairment (creatinine clearance [Cr. Cl.] <50 mL/min, based on Modification of Diet in Renal Disease calculation).
6. Liver function impairment

   1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 × upper limit of normal (ULN), or ALT/AST >3 × ULN plus total bilirubin >2 × ULN.
   2. Total bilirubin >1.5 × ULN, unless the subject has known Gilbert's syndrome.
7. Platelet count <50 000/µL
8. Multi-organ failure.
9. Document active infection with a bacterial pathogen requiring parenteral systemic antibiotics.
10. Bacterial or fungal sepsis.
11. History of live vaccination within the last 4 weeks prior to study enrollment; subjects must not receive live, attenuated influenza vaccine (eg, FluMist) within 4 weeks before enrolment or at any time during the study.
12. History of an allergic reaction or hypersensitivity to the study drug or any component of the study drug formulation.
13. Anti-inflammatory treatments other than steroids (eg, complement inhibitor, anti-GM-CSF antibody, anti-IL6 antibody) ARE PROHIBITED. However, antiviral drugs (eg, remdesivir,), systemic corticosteroids, and non steroidal anti inflammatory drugs (NSAIDs) ARE ALLOWED.
14. Presence of any uncontrolled concomitant illness, serious illness, medical conditions, or other medical history, including laboratory results, which, in the Investigator's opinion, would be likely to interfere with their participation in the study.
15. Major surgical procedure within 4 weeks prior to screening or anticipation of need for major surgical procedure during the course of the study.
16. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to screening
17. History of organ allograft.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with clinical improvement score measured by an 8-point WHO COVID-19 Clinical Improvement Ordinal Scale as assessed by the odds ratio (OR) at Day 14. | at Day 14
  Clinical improvement is defined as
  • A score decrease to categories 1, 2, 3, or 4.

SECONDARY OUTCOMES:
The OR at Days 7, 21, and 28 based on the clinical improvement score (as measured by an 8 point WHO COVID 19 Clinical Improvement Ordinal Scale). | at Day 7, 21, 28
  Clinical improvement defined as per primary endpoint.
The OR at Days 7, 14, 21, and 28 of a decrease of at least 1, 2, 3, and 4 points in subjects with severe COVID 19. | at Day 7, 14, 21, 28
Time to at least 2 point improvement from baseline on Days 7, 14, 21, and 28 in subjects with severe COVID 19. | at Day 7, 14, 21, 28
Worsening (increase in clinical improvement score) of at least '1' score on Days 7, 14, 21, and 28. | at Day 7, 14, 21, 28
Mortality by Days 7, 14, 21, and 28. | up to Day 28
Duration of supplemental oxygen/ventilator support by Days 7, 14, 21, and 28. | up to Day 28
Duration of intensive care unit stay by Days 7, 14, 21, and 28. | up to Day 28
Duration of hospitalization by Days 7, 14, 21, and 28. | up to Day 28
Ventilator free days by Day 14 and Day 28. | up to Day 28
Days on ventilation. | up to Day 28

OTHER OUTCOMES:
Incidence of AEs and treatment-emergent AEs (TEAEs). | up to 28 days
Adverse events leading to premature discontinuation of the study treatment. | up to 28 days
Changes in radiology tests (chest X-ray or chest computed tomography [CT]) from baseline. | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Vuong Trieu, PhD, Study Director — Oncotelic Inc.
Locations (1):
- Praxis Pesquisa Medica S / S Ltda, Jardim, Brazil

IPD SHARING:
Plan to Share IPD: No